CLINICAL TRIAL: NCT00758108
Title: WAGR Syndrome and Other 11p Contiguous Gene Deletions: Clinical Characterization and Correlation With Genotype
Brief Title: Characterization of WAGR Syndrome and Other Chromosome 11 Gene Deletions
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080213; 08-CH-0213
Record Dates: First submitted 2008-09-20; First posted 2008-09-23 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-04-29

CONDITIONS: WAGR Syndrome; Wilm's Tumor; Aniridia; Urogenital Abnormalities; Mental Retardation
Keywords: Genotype/Phenotype Correlation; Energy Homeostasis; Nociception; Obesity; Behavior and Neurocognition; WAGR Syndrome; Wilm's Tumor; Aniridia; Mental Retardation; Urogenital Abnormalities; Healthy Volunteer
MeSH Terms: conditions — WAGR Syndrome; Wilms Tumor; Aniridia; Urogenital Abnormalities; Intellectual Disability; Obesity; Behavior

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will explore conditions caused by the absence of certain genes on chromosome 11. These conditions include WAGR syndrome, which is characterized by a kidney tumor called Wilm s tumor, aniridia (absence of the iris of the eye), genital and urinary abnormalities, mental retardation, and possibly other symptoms. This study will examine how the genes on chromosome 11 affect people and whether the absence of specific genes is associated with specific symptoms.

Healthy normal volunteers, people with isolated aniridia, and people with WAGR or another chromosome 11 gene deletion may be eligible for this study. Participants must be at least 6 years old. Parents of patients may also participate for genetic studies.

Participants undergo some or all of the following procedures, depending on whether they are a child, adult, healthy volunteer or parent of a patient:

* Medical history and physical examination, eye examination, blood, urine and saliva tests, electrocardiogram (EKG) and electroencephalogram (EEG)
* X-rays, scans and other tests to measure body composition (fat, muscle and bone development and thickness) and MRI to examine the eyes and the brain and to measure abdominal fat
* Ultrasound studies of the kidneys, ovaries and uterus (in females) and testes (in males)
* Meal tests, food diaries and food preference tests
* Questionnaires about eating and sleep habits, personality and character traits and responses to pain and injury
* Neuropsychological tests
* Tests of resting metabolic rate, energy expenditure and glucose (sugar) tolerance
* Hot and cold sensitivity tests, vibration sensitivity test, cold tolerance test and smell identification test
* Eye and hearing tests
* Nerve conduction studies and study of sensory information conduction from peripheral nerves to the spinal cord and brain
* Computer photography
* Evaluation by sub-specialists (e.g., endocrinologist, ophthalmologist, physiatrist, neurologist or others) as indicated by the patient s medical history and test results

DETAILED DESCRIPTION:
WAGR syndrome is a rare genetic disorder characterized by Wilms tumor, aniridia, genitourinary anomalies and mental retardation. The syndrome is caused by heterozygous contiguous gene deletions of variable size on chromosome 11, involving a region that encompasses more than 100 genes, many of which have unknown function in humans. In our preliminary studies, we have observed that approximately two-thirds of patients with WAGR syndrome have deletion of the gene which encodes brain-derived neurotrophic factor (BDNF), and that BDNF haploinsufficiency is associated with obesity and with parent reports of hyperphagia and impaired nociception, suggesting that BDNF may play an important role in human energy balance as well as pain sensation. We now propose to conduct a comprehensive clinical phenotype-genotype study on patients with WAGR syndrome and other 11p deletions. We plan to enroll 75 subjects with WAGR syndrome/11p deletions who will undergo evaluations of the following systems: metabolic/endocrine, sensation/nociception, ophthalmologic, audiologic, neurocognitive, renal/genitourinary, oncologic, dental/craniofacial, cardiac, and orthopedic. Genetic testing will be performed on the parents of subjects with WAGR syndrome/11p deletion who choose to participate in order to determine if parental origin of the deletion influences phenotype. We also plan to enroll 75 healthy subjects as body-size matched controls for metabolic studies and 75 patients with isolated aniridia as visually impaired controls for neurocognitive studies. We hypothesize that a more complete understanding of the correlation between phenotype and genotype could lead to improved medical care of these patients through genotype-specific management as well as yield further insight into the physiological role of genes in the 11p region.

ELIGIBILITY:
* INCLUSION CRITERIA:

For WAGR/11p deletion subjects:

1. Diagnosis of WAGR/11p deletion confirmed by prior genetic testing or clinical history consistent with WAGR syndrome (Wilms Tumor and/or genitourinary anomalies plus aniridia). Genetic diagnosis will be confirmed at the NIH, if not done previously
2. Age greater than or equal to 2 years old (Subjects age 2-6y will only have an outpatient evaluation, one 60 mL (or 5 mL/kg if weight <12 kg) blood draw, eye examination, and cognitive, behavioral, and psychiatric assessment performed; subjects age 6y and older will participate in full protocol)
3. Medically stable (so that the patient can safely undergo planned testing); if history of Wilms tumor, must be >6 months since completion of chemotherapy and must be considered in remission by primary oncologist caring for the patient

For parents of WAGR/11p deletion subjects:

a)Biological parent of child with WAGR/11p deletion able to give consent for self participation

For healthy control subjects:

1. Age greater than or eqaul to 2 years old (Subjects age 2-6y will only have an outpatient evaluation, one 60 mL (or 5 mL/kg if weight <12 kg) blood draw, and cognitive, behavioral, and psychiatric assessment performed; subjects age 6y and older will participate in full protocol)
2. No chronic medications. Use of as-needed and over-the-counter medications will be reviewed on a case-by-case basis by the Principal Investigator
3. No chronic medical or psychiatric conditions anticipated to affect results or impede study participation

For aniridia subjects:

1. Diagnosis of aniridia confirmed by ophthalmologist
2. Age greater than or eqaul to 2 years old (Subjects age 2-6y will only have an outpatient evaluation, one 60 mL (or 5 mL/kg if weight <12 kg) blood draw, eye examination, and cognitive, behavioral, and psychiatric assessment performed; subjects age 6y and older will participate in full protocol)
3. Medically stable, with no chronic medical or psychiatric conditions anticipated to affect results or impede study participation

EXCLUSION CRITERIA:

For WAGR/11p deletion subjects:

1. Anorexiant use in preceding 6 months
2. Greater than 2% body weight loss in preceding 6 months
3. Pregnancy
4. Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or other condition which, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study

For parents of WAGR/11p deletion subjects:

a) No exclusions other than lack of ability to give consent for participation

For healthy control subjects:

1. Anorexiant use in preceding 6 months
2. Greater than 2% body weight loss in preceding 6 months
3. Pregnancy
4. Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or other condition which, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study

For aniridia subjects:

1. Anorexiant use in preceding 6 months
2. Greater than 2% body weight loss in preceding 6 months
3. Pregnancy
4. Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or other condition which, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-09-11; Study Completion 2015-04-29

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Breslow NE, Norris R, Norkool PA, Kang T, Beckwith JB, Perlman EJ, Ritchey ML, Green DM, Nichols KE; National Wilms Tumor Study Group. Characteristics and outcomes of children with the Wilms tumor-Aniridia syndrome: a report from the National Wilms Tumor Study Group. J Clin Oncol. 2003 Dec 15;21(24):4579-85. doi: 10.1200/JCO.2003.06.096. PMID 14673045
- [Background] Fischbach BV, Trout KL, Lewis J, Luis CA, Sika M. WAGR syndrome: a clinical review of 54 cases. Pediatrics. 2005 Oct;116(4):984-8. doi: 10.1542/peds.2004-0467. PMID 16199712
- [Background] Pruunsild P, Kazantseva A, Aid T, Palm K, Timmusk T. Dissecting the human BDNF locus: bidirectional transcription, complex splicing, and multiple promoters. Genomics. 2007 Sep;90(3):397-406. doi: 10.1016/j.ygeno.2007.05.004. Epub 2007 Jul 12. PMID 17629449
- [Derived] Sapio MR, Iadarola MJ, LaPaglia DM, Lehky T, Thurm AE, Danley KM, Fuhr SR, Lee MD, Huey AE, Sharp SJ, Tsao JW, Yanovski JA, Mannes AJ, Han JC. Haploinsufficiency of the brain-derived neurotrophic factor gene is associated with reduced pain sensitivity. Pain. 2019 May;160(5):1070-1081. doi: 10.1097/j.pain.0000000000001485. PMID 30855519
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281